CLINICAL TRIAL: NCT05751889
Title: Reducing the Risk of Viral Hepatitis C and Other Sexually Transmitted Infections Among People Living With HIV Who Are Men Who Have Sex With Men: Efficacy of Serious Game Interventions
Brief Title: Serious Game Interventions to Reduce Viral Hepatitis C Among PLWH-MSM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202212073RINC
Record Dates: First submitted 2023-02-09; First posted 2023-03-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Viral Hepatitis C
Keywords: serious game; viral hepatitis C; sexually-transmitted infections; health belief model; harm reduction; sexualized drugs; behavioral interventions
MeSH Terms: conditions — Hepatitis C; Sexually Transmitted Diseases; Harm Reduction

STUDY DESIGN:
Intervention Model Description: Two groups will be assigned to either interventional (serious game intervention) or comparator (traditional health education).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious Game Intervention (Experimental): Provided with a single session serious game intervention regarding HCV and safe sexual practice.
  Interventions: Behavioral: Serious Game
- Traditional Health Education (Active Comparator): Provided with a single session of traditional online healthcare education regarding HCV and safe sexual practice.
  Interventions: Behavioral: Traditional Health Education

INTERVENTIONS:
Behavioral: Serious Game — Serious Game embedded with healthcare information regarding HCV and safe sexual practice.
  Arms: Serious Game Intervention
Behavioral: Traditional Health Education — Reading materials regarding HCV and safe sexual practice.
  Arms: Traditional Health Education

SUMMARY:
The study is aimed to provide high-risk, HIV-infection, men who have sex with men (MSM) with healthcare education regarding viral hepatitis C, through either serious game intervention or traditional online health education. After the education, each participants will be followed for 48 weeks and the change of risky sexual behaviors, acquisition of HCV and other STIs will be followed during the study periods.

DETAILED DESCRIPTION:
High-risk MSM living with HIV were participated in our study will be assigned (by randomization) to either:

1. Serious game intervention: 1 single session of serious game for the participants to play (estimation to take 25-40 minutes). Hepatitis C virus (HCV)-related healthcare informations, including the severity of illness, route of transmission, preventive strategies and treatment options, would be embedded in the game.
2. Traditional online health education (reading materials): 1 single session of healthcare education regarding HCV (with similar contents) will be provided.

After the healthcare intervention, each participants will be followed for 48 weeks. Assessment of risky sexual practice (by questionnaire), test of plasma HCV RNA and serological test of syphilis (optional), and detection of sexually-transmitted bacterial pathogens (optional) will be performed at the enrollment and then every 12 weeks during the observation.

ELIGIBILITY:
Inclusion Criteria:

* High-risk MSM living with HIV, defined as:

  1. Had prior HCV infection, and had cleared HCV through treatment or spontaneously
  2. Had any STI within the past 12 months
  3. Had any unexplained elevation of liver transaminase in the past 6 months
  4. Had at least 1 unprotected anal sex during the past 6 months
* Being able to use mobile smartphone and understand study materials
* Repeat entry of study is permitted, but the interval between health education intervention should >52 weeks.

Exclusion Criteria:

* HCV RNA positive and yet clear virus (nor reaching SVR12).
* Admission for any acute illness (including AIDS-defining conditions)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study targeted MSM living with HIV, which is the major risk group of sexually-transmitted viral hepatitis C in Taiwan.
Enrollment: 1320 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HCV incidence | 48 weeks
  The incidence rate of HCV acquisition between both arms. HCV RNA would be tested for each participants every 3 months during follow-up, and the incidence rate is calculated as following: new cases of HCV viremia / person-time of follow-up.

SECONDARY OUTCOMES:
STI incidence | 48 weeks
  The incidence of sexually-transmitted infection between both arms. Consultation and diagnosis of STI would be performed for each participants every 3 months during follow-up, and the incidence rate is calculated as following: new cases of STI / person-time of follow-up.
The frequency of condom use and sexualized drug use | At weeks 12, 24 and 48 of observation
  The frequency engaging in condomless sex and the use of sexualized drugs (within the past 3 months) will be assessed for each participant at the enrollment, week 12, 24 , and 48. We would compare the change these behaviors at week 12, 24 and 48 to the baseline to see if there are difference between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
However, de-identified data regarding the pre-defined outcomes or relevant characteristics could be available per request.